CLINICAL TRIAL: NCT04006262
Title: Peri-operative Association of Immunotherapy (Pre-operative Association of Nivolumab and Ipilimumab, Post-operative Nivolumab Alone) in Localized Microsatellite Instability (MSI) and/or Deficient Mismatch Repair (dMMR) Oeso-gastric Adenocarcinoma: An Open-label GERCOR Phase II Study
Brief Title: Pre-operative Nivolumab and Ipilimumab, Followed by Post-operative Nivolumab, for MSI/dMMR Oeso-gastric Adenocarcinoma.
Acronym: NEONIPIGA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEONIPIGA - D18-02
Record Dates: First submitted 2019-06-17; First posted 2019-07-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Localized Oesogastric Adenocarcimona; MSI and or dMMR
MeSH Terms: conditions — Microsatellite Instability | interventions — Nivolumab; Ipilimumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): * Neo-adjuvant treatment (6 cycles - 12 weeks)
  * Surgery
  * Adjuvant treatment (9 cycles - 9 months)
  Interventions: Drug: Nivolumab 10 MG/ML; Drug: Ipilimumab 200 MG in 40 ML Injection

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML — Neo-adjuvant treatment : 240 mg intravenous (I.V.) in 30 minutes - every 2 weeks - 6 cycles
  - Adjuvant treatment : 480mg I.V. in 30 minutes - every 4 weeks - 9 cycles
  Other Names: Opdivo
Drug: Ipilimumab 200 MG in 40 ML Injection — Neo-adjuvant treatment : 1mg/kg over 30 minutes every 6 cycles - 2 cycles
  Other Names: Yervoy

SUMMARY:
This is a non-randomized study, open label phase II study. The purpose of this study is to evaluate the complete pathologic response rate (cPRR) with neoadjuvant nivolumab and ipilimumab combination in patients with MSI and/or dMMR localized oeso-gastric cancer.

DETAILED DESCRIPTION:
In patients with resectable oeso-gastric adenocarcinoma, radical surgery is the only curative option. Despite the evolution in treatment with multimodality treatment strategies, oeso-gastric cancer remains one of the most lethal malignancies with 5-year survival rates reaching only 22%. When the disease is localized, perioperative chemotherapy with cytotoxic agents is the preferred strategy since it increases the overall survival (OS) rate. However, in oeso-gastric cancers with microsatellite instability (MSI), is a favorable prognostic factor, the recommended cytotoxic chemotherapy combination seems inefficient and even deleterious.

It is now well established that dMMR and or the MSI phenotype are the surrogate markers of response to immunotherapy.

The combination of nivolumab and ipilimumab had shown promising efficacy in multiple tumor types (dMMR/MSI).

Based on the data above, we have designed this phase II study to evaluate the complete pathological response rate (cPRR) in patients with non-metastatic MSI/dMMR oeso-gastric adenocarcinoma treated with neoadjuvant nivolumab and ipilimumab treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent,
2. Age ≥18 years to ≤75 years of age,
3. Histologically proven non-metastatic gastric adenocarcinoma or of the oeso-gastric junction T2 to T4, Nx, M0 after thoraco-abdominopelvic computed tomography (CT) and echo-endoscopy,
4. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study,
5. dMMR (protein expression by immunohistochemistry [ICH] and/or MSI by polymerase chain reaction [PCR]), MMR and/or MSI tumors should be assessed per local guidelines: ICH with two (anti-MLH1 and anti-MSH2 or anti-MSH6, and antiPMS2) or four antibodies (anti-MLH1, anti-MSH2, anti-MSH6, and anti-PMS2) and/or PCR (with PROMEGA: BAT- 25, BAT-26, NR-21, NR-24, and NR-27) by the investigators prior to screening, Extinct MLH1 (+/- PMS2), MSH2 (+/- MSH6), MSH6, or PMS2 alone protein expression by IHC (dMMR), and/or tumor with ≥ 2 instable MSI-H markers on PCR: BAT25, BAT26, NR21, NR24, and NR27 (pentaplex panel is recommended),
6. The Eastern Cooperative Oncology Group Performance status (ECOG PS) 0-1, for patients over 70 years ECOG PS of 0;
7. Hematological status: absolute neutrophil count (ANC) ≥1.5 x 109/L; platelets ≥100 x 109/L; hemoglobin ≥9 g/dL,
8. Adequate renal function: serum creatinine level <120 µM, clearance > 50ml/min (Modification of the Diet in Renal Disease [MDRD] or Cockcroft and Gault),
9. Adequate liver function: serum bilirubin ≤1.5 x upper normal limit (ULN), alkaline phosphatase <5 x ULN, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤3.0 x ULN,
10. No prior therapy for localized oeso-gastric cancer,
11. Radiological tumor assessment within 21 days before the start of treatment according to RECIST version 1.1 by Chest Abdomen and Pelvis CT,
12. For female patients of childbearing potential, negative pregnancy test within 7 days before starting the study drug,
13. Men and women are required to use adequate birth control during the study (when applicable), Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use a highly effective method of birth control (i.e., pregnancy rate of less than 1% per year) during the period of treatment and during 5 and 7 months, woman and men, respectively, from the last treatment administration. Men must refrain from donating sperm during this same period, Contraceptive methods that result in a low failure rate when used consistently and correctly include methods such as combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), some intrauterine devices, intrauterine hormone- releasing stem, true sexual abstinence (when this is in line with the preferred and usual lifestyle of the participant), bilateral tubal occlusion, or a female partner who is not of childbearing potential or a male partner who has had a vasectomy. Women and female partners using hormonal contraceptive must also use a barrier method i.e. condom or occlusive cap (diaphragm or cervical/vault caps), A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus),
14. Subject willing to comply to provide primary tumor tissue (archival or fresh biopsy specimen), including possible pre-treatment biopsy for PD-L1 expression analysis and other biomarker correlative studies
15. Registration in a National Health Care System (PUMa - Protection Universelle Maladie included)

Exclusion Criteria:

Non-eligible to clinical trial if one of following parameter is reported:

1. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
2. Treatment with any investigational medicinal product within 28 days prior to study entry,
3. Major surgical procedure within 4 weeks prior to initiation of study treatment,
4. Other serious and uncontrolled non-malignant disease (including active infection),
5. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
6. Metastases (M stage disease) whatever the location,
7. Pregnant or breastfeeding women,
8. Human immunodeficiency virus (HIV),
9. Active hepatitis B virus (HBV, defined as having a positive hepatitis B surface antigen [HBsAg] test prior to inclusion) or hepatitis C virus (HCV). Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible. Note: Patients positive for HCV antibody are eligible only if PCR testing is negative for HCV RNA
10. Patient on tutelage or guardianship or under the protection of justice.
11. Impossibility of submitting to the medical follow-up of the study for geographical, social or psychiatric reasons.

Non-eligible to immunotherapy:

1. History of autoimmune disease including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, Note: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible. Note: Controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
2. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest imaging,
3. Administration of a live, attenuated vaccine within 4 weeks prior to start of treatment or anticipation that such a live attenuated vaccine will be required during the remainder of the study,
4. Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or antiPD-L1 therapeutic antibody or pathway-targeting agents,
5. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
6. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including, but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to start of adjuvant treatment, or requirement for systemic immunosuppressive medications during the remainder of the study. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Note: Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled into the study after approval of the Medical Contact. Subjects are permitted the use of topical, ocular, intra- articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).

Adrenal replacement steroid doses including doses >10 mg daily prednisone is permitted. A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g. contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by a contact allergen) is permitted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Complete pathological response (cPRR) rate | time point when the tumor is examined after the surgery (up to 30 months)
  Each center will assess the pathologic response with a centralized center review in case of cPRR and the analysis will be in intention-to-treat (ITT).
  cPRR will be defined as complete tumor disappearance of tumor in the low esophagus or the stomach (from 1/3 inferior of the esophagus to pylorus) after surgery anatomopathologic examination according to mandard scale.
  Surgery will be performed within 5 weeks +\- 1 week after the last cycle (cycle 6) of neoadjuvant therapy

SECONDARY OUTCOMES:
Disease-free survival (DFS) | Up to 36 months
  DFS is defined as the time from the date of starting treatment to local recurrence and/or metastases or death irrespective of cause and censored at the date of last contact.
Overall Survival (OS) | Up to 36 months
  OS is defined as the time between the date of the first dose of study treatment and the death date. Patients alive at last report will be considered censored at the endpoint. Alive patients will be censored at the last date known to be alive, either during study treatment period or during follow-up period.
Number of participants with treatment-related adverse events | Patients will be assessed for AEs throughout the study at every visit during treatment and at 3-month follow-up visit (3 months after treatment ends). Investigators using the NCI-CTCAE version 5.0 will grade the severity of AEs.
  Number of participants with treatment-related adverse events as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v5.0
Analyze MSI status | up to 36 months
  Confirmation of MSI and/or dMMR has to be confirmed retrospectively on archival or fresh tumor FFPET block from the primary tumor obtained at the time of the initial diagnosis
Quantification of antigen-specific CD4+ T cells as biomarker of anti-PD1/PDL1 immunotherapy in dMMR tumors | Blood samples at baseline, C3D1 and C6D1 of neoadjuvant therapy - cycle every 2 weeks, after surgery at C1 D1(first cycle of adjuvant treatment) and at the end of treatment visit (28 days after the last dose of treatment (up to 36 months)
  Quantification of antigen-specific CD4+ T cells as biomarker of anti-PD1/PDL1 immunotherapy in blood of dMMR tumors.
Number of Species of bacteria and yeast composition | Baseline and at week 12
  To investigate the microbiota composition changes during neoadjuvant therapy with nivolumab and ipilimumab and its relation to response and/or chemotoxicity.
  Number of Species of bacteria and yeast will be quantitfy and identify. Number of Change of composition will be investigate based on baseline samples compared to 12 weeks sample.
  DNA will be extracted from fecal samples taken prior to therapy and on-treatment (week 12). A gene sequencing approach will be utilized to survey microbial species in the gut in order to define microbiota as a function of the efficacy and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry ANDRE, MD, Principal Investigator — Hôpital Saint Antoine PARIS
Locations (15):
- France (15):
  - CHRU Jean Minjoz, Besançon
  - Hôpital Henri Mondor, Créteil
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - CHRU Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - ICM Val d'Aurelle, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Européen Geroges Pompidou, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - CHU Pontchaillou Rennes, Rennes
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andre T, Tougeron D, Piessen G, de la Fouchardiere C, Louvet C, Adenis A, Jary M, Tournigand C, Aparicio T, Desrame J, Lievre A, Garcia-Larnicol ML, Pudlarz T, Cohen R, Memmi S, Vernerey D, Henriques J, Lefevre JH, Svrcek M. Neoadjuvant Nivolumab Plus Ipilimumab and Adjuvant Nivolumab in Localized Deficient Mismatch Repair/Microsatellite Instability-High Gastric or Esophagogastric Junction Adenocarcinoma: The GERCOR NEONIPIGA Phase II Study. J Clin Oncol. 2023 Jan 10;41(2):255-265. doi: 10.1200/JCO.22.00686. Epub 2022 Aug 15. PMID 35969830